CLINICAL TRIAL: NCT00838006
Title: Identification of and At-Risk Interventions for Pre-deployment Psychophysiologic Predictors of Post-deployment Mental Health Outcomes
Brief Title: Psychophysiologic Predictors of Post-deployment Mental Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biomedical Research Foundation (Other)
Responsible Party: Principal Investigator, Jeffrey Pyne, Research Scientist, Biomedical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PT074626
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Post-traumatic Stress Disorder
Keywords: post-traumatic stress disorder; post-deployment; prediction; prevention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biofeedback training (Experimental): Heart rate variability biofeedback training and iPod with Breath Pacer app
  Interventions: Device: heart rate variability biofeedback
- Cognitive bias modification training (Experimental): Cognitive bias modification training and iPod with cognitive bias training app
  Interventions: Device: Cognitive bias modification training
- Control Group (Sham Comparator): No additional resilience training and iPod with no resilience training apps
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: heart rate variability biofeedback — Heart rate variability biofeedback, 3 session plus handheld device
  Arms: Biofeedback training
Device: Cognitive bias modification training — Cognitive bias modification training - 3 session plus handheld device
  Arms: Cognitive bias modification training
Device: Sham Comparator — Subjects received iPod without a study app and no additional resilience training
  Arms: Control Group

SUMMARY:
The primary objectives of this proposal are to develop objective pre-deployment predictors of PTSD and test two pre-deployment resiliency interventions.

DETAILED DESCRIPTION:
The primary objectives of this proposal are to develop objective pre-deployment predictors of PTSD and test two pre-deployment resiliency interventions. The objective predictors will be based on: 1) physiologic reactivity (heart rate, heart rate variability, eye blink startle, skin conductance) to virtual reality (VR) environments depicting common Operation Iraqi Freedom (OIF) or Operation Enduring Freedom (OEF) combat scenarios and 2) cognitive bias assessment using a recognition memory paradigm. We hypothesize that a model combining physiologic reactivity and cognitive bias predictors will be superior to either the physiologic reactivity or cognitive bias model alone for predicting post-deployment PTSD. We also will test two pre-deployment resiliency interventions: heart rate variability biofeedback and cognitive bias modification training that we have designed to target physiologic and cognitive responses to stress, respectively. We will compare the prevention interventions to a no intervention control group. We hypothesize that the prevalence of post-deployment PTSD will be lower in the intervention groups compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Army National Guard members who are scheduled to deploy for OIF/OEF operations within the next 12 months, age 18 to 60, and willing to provide the name and phone number of at least one person to help locate the member for the follow-up assessments if necessary.

Exclusion Criteria:

* Implantable pacemaker or cardiac defibrillator
* Unable to wear a virtual reality headset

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 426 (Actual)
Dates: Start 2008-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Pyne, MD, Principal Investigator — Central Arkansas Veterans Healthcare System
Locations (1):
- Virginia Army National Guard, Blackstone, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 426 soldiers were enrolled and completed the pre-deployment assessment. Fo these, 342 were randomized and had at least one follow-up assessment.
Groups:
- Heart Rate Variability Biofeedback Training: Heart rate variability biofeedback training and iPod with Breath Pacer app
  heart rate variability biofeedback: Heart rate variability biofeedback,1 session plus handheld device
- Cognitive Bias Modification Training: Cognitive bias modification training and iPod with cognitive bias training app
  Cognitive bias modification training: Cognitive bias modification training - 1 session plus handheld device
Period: Overall Study
Arm/Group | Heart Rate Variability Biofeedback Training | Cognitive Bias Modification Training | Control Group
Started | 102 | 98 | 142
3-month Post-deployment Follow-up | 92 | 80 | 135
Completed | 68 | 72 | 94
Not Completed | 34 | 26 | 48

BASELINE CHARACTERISTICS:
Population: 342 participants completed at least one follow-up and were included in the analysis
Groups:
- Cognitive Bias Modification: Soldiers randomized to Cognitive Bias Modification for Interpretation training arm
- Heart Rate Variability Biofeedback: Soldiers randomized to Heart Rate Variability Biofeedback training arm
- Control: Soldiers randomly assigned to Control group
- Total: Total of all reporting groups
Arm/Group | Cognitive Bias Modification | Heart Rate Variability Biofeedback | Control | Total
Number analyzed (Participants) | 98 | 102 | 142 | 342
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 98 | 102 | 142 | 342
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (8.5) | 29.0 (8.6) | 28.1 (8.2) | 28.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 16 | 6 | 28
  Male | 92 | 86 | 136 | 314
Region of Enrollment [Number; unit: participants]
  United States | 98 | 102 | 142 | 342

OUTCOME MEASURES:

1. Primary Outcome: The PTSD Checklist - Military Version
Description: The Post Traumatic Stress Disorder Checklist is based on Diagnostic Statistical Manual (DSM)-IV symptoms of PTSD. The minimum score is 17 and the maximum score is 85. Higher scores are associated with more severe symptoms and worse outcome.
Time Frame: pre-deployment, 3-, and 12-months post-deployment
Population: participants completed baseline and at least one follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- HRV Biofeedback: Soldiers randomized the heart rate variability biofeedback training arm
- Cognitive Bias Modification Training: Soldiers randomized to the cognitive bias modification for interpretation training arm
- Control: Soldiers randomized to the control arm
Arm/Group | HRV Biofeedback | Cognitive Bias Modification Training | Control
Number analyzed (Participants) | 102 | 98 | 142
units on a scale
  Pre-deployment | 22.2 (6.6) | 23.7 (8.4) | 23.8 (9.6)
  3-months Post-deployment | 25.9 (9.2) | 26.5 (11.9) | 28.5 (12.7)
  12-month Post-deployment | 24.5 (9.2) | 24.3 (8.6) | 23.9 (9.7)

2. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 is a nine-item depression module that is based on DSM-IV criteria for major depression. The minimum score is 0 and the maximum score is 27. Higher scores indicate more severe depression or worse outcome.
Time Frame: pre-deployment, 3-, and 12-month post-deployment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Heart Rate Variability Biofeedback Training: Soldiers randomized the heart rate variability biofeedback training arm
Arm/Group | Heart Rate Variability Biofeedback Training | Cognitive Bias Modification Training | Control
Number analyzed (Participants) | 102 | 98 | 142
units on a scale | 2.83 (3.19) | 3.02 (3.27) | 3.03 (3.29)

ADVERSE EVENTS:
Groups:
- HRV Biofeedback: Soldiers randomized to heart rate variability biofeedback training arm
- Cognitive Bias Modification Training: Soldiers randomized to Cognitive Bias Modification for Interpretation training arm
Arm/Group | HRV Biofeedback | Cognitive Bias Modification Training | Control
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/98 | 0/142
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/98 | 0/142
Other Adverse Events (participants affected / at risk) | 0/102 | 0/98 | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No